CLINICAL TRIAL: NCT02577562
Title: Zenith® Fenestrated AAA Endovascular Graft Clinical Study
Brief Title: Zenith® Fenestrated Abdominal Aortic Aneurysm (AAA) Endovascular Graft Continued Access Study
Status: Approved for marketing | Type: Expanded Access
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 04-541 CA
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Abdominal Aortic Aneurysms; Aorto-iliac Aneurysms; Juxtarenal Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

INTERVENTIONS:
Device: Zenith® Fenestrated AAA Endovascular Graft — The Zenith® Fenestrated AAA Endovascular Graft with the H&L-B One-Shot™ Introduction System is indicated for the endovascular treatment of patients with abdominal aortic or aortoiliac aneurysms having morphology suitable for endovascular repair

SUMMARY:
The Zenith®Fenestrated AAA Endovascular Graft Clinical Study is a clinical investigation approved by the US FDA to study the safety and effectiveness of the Zenith® Fenestrated AAA Endovascular Graft in the treatment of abdominal aortic and aorto-iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic and aortoiliac aneurysms with diameter greater than or equal to 5 cm

Exclusion Criteria:

* Proximal neck less than 4 mm or greater than or equal to 15 mm in length unless otherwise compromised to preclude seal
* Renal artery stenosis greater than 50 percent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of California, San Francisco, San Francisco, California
  - Shands Hospital, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Medical Center, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Harborview Medical Center, Seattle, Washington